CLINICAL TRIAL: NCT05946850
Title: Caudal Analgesia in Anticoagulated Chronic Pain Patients
Brief Title: Caudal Analgesia & Anticoagulated Patient
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Salem2018 Caudal Blk Anticoag
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Pain Syndrome; Anticoagulants and Bleeding Disorders
Keywords: Caudal analgesia
MeSH Terms: conditions — Somatoform Disorders; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Caudal analgesia — Caudal analgesia for chronic lumbosacral pain

SUMMARY:
Caudal analgesia is an effective intervention for lumbosacral pain. Some chronic pain patients take anticoagulants for vasculopathy treatment. Anticoagulation limits the use of caudal analgesia because of the risk of epidural bleeding. Caudal analgesia may be safe and effective in anticoagulated chronic pain patients.

Quantitative analysis of prospective clinical data. Evaluation of caudal analgesia efficacy and safety in anticoagulated chronic pain patients. Analysis of outcome, and complications.

DETAILED DESCRIPTION:
Caudal analgesia is an effective interventional therapy for chronic lumbosacral pain. Some chronic pain patients take anticoagulants for vasculopathy treatment. Anticoagulation limits the use of caudal analgesia because of the risk of epidural bleeding. Anticoagulation may be discontinued briefly, to allow caudal injection. Interruption of anticoagulation may be difficult and dangerous for some high-risk patients. Caudal analgesia may be safe and effective in anticoagulated chronic pain patients.

Quantitative analysis of prospective clinical data. An evaluation of caudal analgesia safety in anticoagulated chronic pain patients. An analysis of treatment outcome, and complications.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients who undergo caudal analgesia

Exclusion Criteria:

* chronic pain patients who refuse caudal analgesia

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain clinic patients who have lumbosacral pain, and undergo caudal analgesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 12 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Boswell MV, Singh V, Benyamin RM, Fellows B, Abdi S, Buenaventura RM, Conn A, Datta S, Derby R, Falco FJ, Erhart S, Diwan S, Hayek SM, Helm S, Parr AT, Schultz DM, Smith HS, Wolfer LR, Hirsch JA; ASIPP-IPM. Comprehensive evidence-based guidelines for interventional techniques in the management of chronic spinal pain. Pain Physician. 2009 Jul-Aug;12(4):699-802. PMID 19644537